CLINICAL TRIAL: NCT05213143
Title: The Safety and Efficacy of Lurasidone In Subjects With Schizophrenia Switched From Olanzapine: An Open-label, Single-arm And Multi-center Study for 16 Weeks
Brief Title: The Safety and Efficacy of Lurasidone In Subjects With Schizophrenia Switched From Olanzapine
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Company's business decision
Sponsor: Sumitomo Pharma (Suzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DSPC-LAT-002
Record Dates: First submitted 2021-12-05; First posted 2022-01-28 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Lurasidone Hydrochloride

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Lurasidone (Experimental): Lurasidone was oral administrated with a meal or within 30 min after eating in the evening.
  Interventions: Drug: Lurasidone

INTERVENTIONS:
Drug: Lurasidone — Lurasidone was oral administrated with a meal or within 30 min after eating in the evening. The maintenance dose of olanzapine from Day 0 to Day 6, than tapered until discontinuation from Day 7 to Day 27. Lurasidone initiated with 40mg/d on Day 0, maintained until Day 13, with a flexible dose (40-80mg/d, qd) from Day 28 to Day 111.

SUMMARY:
An open-label, single-arm and multi-center study for 16 weeks

DETAILED DESCRIPTION:
An open-label, single-arm and multi-center study for 16 weeks, to study the improvement of weight gain in patients with schizophrenia who switched from olanzapine to lurasidone.

ELIGIBILITY:
Inclusion Criteria:

* Subject aged ≥ 18 to ≤ 65 years old
* Meet ICD-10 criteria for a primary diagnosis of schizophrenia， the duration must be at least one year
* Provide written informed consent (subject's legal guardian or impartial witness shall sign informed consent if the subject is unable to sign) and is willing and able to comply with the protocol in the opinion of the investigator.
* Considered to be an appropriate candidate for switching olanzapine due to safety or tolerability concerns
* Received Olanzapine monotherapy at a dose of 10 to 20mg/d for at least 8 weeks with a body mass index (BMI) ≥25kg/m2, the dose of olanzapine has been stable for at least 4 weeks prior to screening. Weight gain during current olanzapine therapy was verified in the subject history.
* Subject must meet the clinical stability as following criteria:

  1. CGI-S ≤ 4 (at both Screening and Baseline)
  2. PANSS total score ≤ 70 at Screening and Baseline
  3. No exacerbation of schizophrenia has occurred for at least 8 weeks prior to screening

Exclusion Criteria:

* Subjects with severe or unstable physical diseases (including but not limited to severe or unstable cardiovascular diseases, cerebrovascular diseases, liver and kidney diseases) determined by the investigators.
* Currently has severe liver function impairment, or serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) level ≥3 times the upper limit of normal value
* Creatinine clearance rate < 50mL/min
* Subjects had a history of stomach or intestinal surgery or any other condition that could interfere with absorption, distribution, metabolism, or excretion of medications
* More than 10% weight loss 3 months prior to the screening period
* A history of malignant tumors (including benign pituitary tumors)
* Any chronic organic disease of the central nervous system (excluding schizophrenia), such as CNS related tumors and inflammation, active seizures, vascular disease, Parkinson's disease, Alzheimer's disease, or other forms of dementia, myasthenia gravis, and other degenerative diseases. A history of mental retardation or persistent neurological symptoms caused by severe head injury
* Subjects need to take any potent CYP3A4 inhibitor (e.g., ketoconazole, ritonavir, clarithromycin, ritonavir, voriconazole, Mibefradil) or inducer (e.g. rifampicin, avasimibe, St. John's Wort, phenytoin, carbamazepine), drugs for external use in dermatological patients are excluded
* Subject has a history of treatment with clozapine for refractory psychosis and/or subject has been treated with clozapine (for any reason) within 4 months of baseline
* Subjects has used long-term antipsychotic drugs in the following time prior to the enrolment
* Subjects received electroconvulsive therapy (ECT) within 90 days prior to screening, or were expected to require ECT during the study
* A history of neuroleptic malignant syndrome
* Severe tardive dyskinesia, severe dystonia, or any other severe dyskinesia
* Subjects is at risk of suicide or self-mutilation behaviours or the act of endangering others, or other corresponding characteristic behaviour, or a history of suicide
* Female subjects were pregnant (positive pregnancy test at screening) or breast-feeding or planning pregnancy for the duration of the study, or the partners of male subjects were planning pregnancy for the duration of the study
* History of severe allergy or hypersensitivity;
* Angioedema occurred after previous administration of lurasidone;
* Patients who had previously participated in a clinical study of lurasidone;
* The subject is participating in or has participated in other clinical trials, including the use of commercially available drugs or medical devices, within 30 days prior to the signing of the informed consent;
* Any other conditions judged by the investigators that not suitable to participate in this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-12-30 (Actual); Primary Completion 2022-11-18 (Actual); Study Completion 2022-11-18 (Actual)

PRIMARY OUTCOMES:
Mean weight change | from baseline to week 16
  Changes in body weight at the end of treatment compared to baseline

SECONDARY OUTCOMES:
Change in Positive and Negative Syndrome Scale (PANSS) scores | from baseline to week 16
  Change in PANSS scores at the end of treatment compared to baseline.
Change in the Clinical Global Impressions-Severity (CGI-S) scores | from baseline to week 16
  Change in CGI-S scores at the end of treatment compared to baseline.
Change in 12-Item Short Form Survey (SF-12) scores | from baseline to week 16
  Change in SF-12 scores at the end of treatment compared to baseline
Change in waist circumference | from baseline to week 16
  Change in waist circumference at the end of treatment compared to baseline. Wrap the tape around 0.5 to 1.0 cm above the belly button, and measure the circumference.Obese patients wrap a tape measure around the widest part of their waist.
Change in the serum prolactin (PRL) | from baseline to week 16
  Change in PRL at the end of treatment compared to baseline.
Change in Calgary Depression Scale for Schizophrenia (CDSS) scores | from baseline to week 16
  Change in CDSS scores at the end of treatment compared to baseline.
Change in fasting lipids | from baseline to week 16
  Change in fasting lipids（total cholesterol, triglycerides, high density liptein cholesterol, low density lipoprotein, Non-high density liptein cholesterol) at the end of treatment compared to baseline.
Change in fasting plasma glucose | from baseline to week 16
  Change in fasting plasma glucose at the end of treatment compared to baseline.
Change in hemoglobin A1c (HbA1c) | from baseline to week 16
  Change in HbA1c at the end of treatment compared to baseline.
Change in the Epworth Sleepiness Scale | from baseline to week 16
  Change in the Epworth sleepiness scale at the end of treatment compared to baseline. A score of 10 or greater raises concern.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anding Hospital, Beijing, Beijing Municipality, China